CLINICAL TRIAL: NCT06695949
Title: Comparison of Percutaneous Neuromodulation and Therapeutic Exercise in Patients With Nonspecific Chronic Neck Pain: A Randomized Clinical Trial
Brief Title: Percutaneous Neuromodulation and Therapeutic Exercise in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, Full Profesor, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP-0429-2023-C4
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neck Pain; Chronic Pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous neuromodulation (Experimental): Patients assigned to this group (n=50) will receive one weekly sessions of percutaneous neuromodulation for a total of 6 weeks, with each session lasting 30 minutes. For the treatment application, the patient will be positioned in a prone decubitus position, leaving the dorsal-cervical area exposed, and we will apply skin disinfectant (chlorhexidine). Subsequently, and under ultrasound guidance, we will perform the technique using a 30 x 40 mm acupuncture needle, which will be inserted at three vertebral levels and bilaterally: the greater occipital nerve (C0-C1), and the posterior roots of vertebral levels C3-C4 and C7-T1, the spinal nerve, suprascapular nerve and dorsal. Once the needles are correctly positioned, we will connect alligator clip electrodes segmentally, connecting them to an electrotherapy device (TensMed S82-Enraf Nonius) applying a TENS current. The parameters used will be set to low-frequency (2 Hz) symmetric biphasic pulsed current with a pulse width of 120 μs
  Interventions: Other: Percutaneous neuromodulation.
- Therapeutic Exercise (Other): These participants (n=50) will engage in resistance training for the cervical flexor muscles, following a progressive exercise program in a supine position with the head comfortably supported, as described by Falla et al. (2008). Participants will perform these exercises with a frequency of 3 days a week for 6 weeks, with each session lasting 30 minutes.
  Interventions: Other: Therapeutic Exercise.

INTERVENTIONS:
Other: Percutaneous neuromodulation. — Percutaneous neuromodulation therapy involves inserting several fine needle electrodes 2 cm to 5 cm deep into the skin to target the muscle and surrounding soft tissues. A low-voltage electric current is then passed through these needles, which is hypothesized to improve muscle function by altering the pain signals traveling from the painful muscle to the brain, enhance blood flow to the painful area to promote healing, reduce inflammation and soreness, and increase muscle endurance, strength, and balance.
  Other Names: Experimental
  Arms: Percutaneous neuromodulation
Other: Therapeutic Exercise. — These participants (n=50) will engage in resistance training for the cervical flexor muscles, following a progressive exercise program in a supine position with the head comfortably supported, as described by Falla et al. (2008). Participants will perform these exercises with a frequency of 3 days a week for 6 weeks, with each session lasting 30 minutes.
  Other Names: Active Comparator
  Arms: Therapeutic Exercise

SUMMARY:
The aim of this study is to compare the effects of applying percutaneous neuromodulation with performing only therapeutic exercise in patients with non-specific chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is highly prevalent, affecting 203 million people worldwide in 2020 and ranking eleventh in terms of years lived with disability. More than 50% of individuals will not recover from an acute episode and will experience recurrent neck pain within 1 to 5 years, leading to a persistent and chronic problem. Chronic neck pain can originate from a traumatic episode, such as whiplash, or it may not have a traumatic origin. In the latter case, in the absence of an identifiable pathoanatomic cause, it is classified as nonspecific chronic neck pain (NSNP). The GBD 2021 study acknowledges that the burden of neck pain has not been reduced in the past three decades and projects a significant increase in this absolute burden by 2050. Several studies have highlighted the urgency of prioritizing future research on preventing and treating this condition.

Clinical practice guidelines for the management of NSNP advocate for the use of exercise. Specifically, it has been shown that specific neck exercises are more effective than other types of alternative exercises in reducing pain and disability in patients with NSNP. In recent years, treatment based on percutaneous neuromodulation (PNM) has gained popularity and has become an alternative to conventional treatment for soft tissue injuries, noted for its low incidence of significant side effects. PNM involves the percutaneous electrical stimulation of a peripheral nerve, either along its pathway or in a muscle, using a puncture needle that utilizes low or medium-frequency electrical currents. Additionally, the advent of ultrasound technology has provided new opportunities to improve the safety of this invasive approach.

The primary goal of PNM is to relieve pain and restore the normal functioning of the nervous system, reducing chronic and neuropathic pain associated with central sensitization and improving neuromuscular function and motor control. Although the physiological mechanism explaining pain inhibition and the analgesic effect remains incomplete, various hypotheses have been proposed to expand current knowledge. Among the most cited models is the "gate control" theory, which suggests that the electrical stimulation of large-diameter afferent nerve fibers inhibits pain transmission through small-diameter fibers to the central nervous system at the spinal cord level, producing what is known as neuromodulation. However, few studies investigate the effects of PNM, so more evidence is needed to draw solid conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 30 and 65 years with chronic cervical pain.
* Chronic cervical pain lasting 3 months or more and not receiving any other type of physiotherapy treatment.

Exclusion Criteria:

* Patients with sensory and/or coagulation disorders.
* History of spine surgery, cardiac complications, and severe concurrent central or peripheral nervous system disease.
* Epilepsy, needle phobia, disc pathology, or serious pathologies that may be the primary cause of chronic cervical pain (e.g., tumors, Arnold Chiari disease, vertigo syndrome, etc.)
* Contraindications for transcutaneous electrical nerve stimulation (TENS).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Neck disability index | At baseline, at 6 weeks and at 8 weekss.
  The neck disability index consists of 10 questions addressing functional activities such as personal care, lifting, reading, work, driving, sleeping, recreational, pain intensity, concentration and headache.
Pain (Visual Analog Scale) | At baseline, at 6 weeks and at 8 weeks.
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).

SECONDARY OUTCOMES:
Pain (Visual Analog Scale) | At baseline, at 6 weeks and at 8 weeks.
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
McGill Pain Questionnaire | At baseline, at 6 weeks and at 8 weeks.
  The McGill Pain Questionnaire is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. The MPQ is a multi-dimesional tool for pain assessment and it has three components, which are the sensory intensity, the cognitive evaluation of pain and the emotional impact of pain.
Quality of Life (SF-36 quality of life questionnaire) | At baseline, at 6 weeks and at 8 weeks.
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
Quality of Sleep (Pittsburgh Quality of Sleep Questionnaire Index) | At baseline, at 6 weeks and at 8 weeks.
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction.
Tampa scale for kinesiophobia | At baseline, at 6 weeks and at 8 weeks.
  The 17-item Tampa scale for kinesiophobia assesses fear of movement or of injury or reinjury.
Pain Catastrophizing Scale | At baseline, at 6 weeks and at 8 weeks.
  The Pain Catastrophizing Scale (PCS) is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. Catastrophizing is commonly described as an exaggerated negative orientation toward noxious stimuli and plays an important role in experiencing and coping with pain. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale.
Treatment expectations | At baseline, at 6 weeks and at 8 weeks.
  Questionnaire on treatment expectations and the patient's perception level
Expectations regarding cervical pain | At baseline, at 6 weeks and at 8 weeks.
  Questionnaire on expectations regarding cervical pain.
Cervical Range of Motion (Pro Motion Capture. Werium) | At baseline, at 6 weeks and at 8 weeks.
  Cervical range of motion is assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90º of flexion, and buttocks positioned against the back of the chair.
Active and Latent Myofascial Trigger Points (Number of trigger Points) | At baseline, at 6 weeks and at 8 weeks.
  Myofascial Trigger Points will be explored in the following pairs of muscles: occipitofrontalis, splenius capitis, sternocleidomastoid, anterior scalene, middle scalene, posterior scalene, upper trapezius, middle trapezius, lower trapezius, supraspinatus, infraspinatus, and multifidus level C6.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida María Castro-Sánchez, PhD, Principal Investigator — Universidad de Almeria
Locations (1):
- University of Almeria, Almería, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study data will be available by email at ilp813@ual, provided that a reasonable request is made with justification for its scientific use and that citation is guaranteed.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning with the first article publication; ending 5 years following article publication.
Access Criteria: Data will be accessed via the contact email ilp813@ual.es, provided that its scientific use and citation of our protocol are guaranteed.

REFERENCES:
- [Background] Kazeminasab S, Nejadghaderi SA, Amiri P, Pourfathi H, Araj-Khodaei M, Sullman MJM, Kolahi AA, Safiri S. Neck pain: global epidemiology, trends and risk factors. BMC Musculoskelet Disord. 2022 Jan 3;23(1):26. doi: 10.1186/s12891-021-04957-4. PMID 34980079
- [Background] GBD 2021 Neck Pain Collaborators. Global, regional, and national burden of neck pain, 1990-2020, and projections to 2050: a systematic analysis of the Global Burden of Disease Study 2021. Lancet Rheumatol. 2024 Mar;6(3):e142-e155. doi: 10.1016/S2665-9913(23)00321-1. PMID 38383088
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Fandim JV, Nitzsche R, Michaleff ZA, Pena Costa LO, Saragiotto B. The contemporary management of neck pain in adults. Pain Manag. 2021 Jan;11(1):75-87. doi: 10.2217/pmt-2020-0046. Epub 2020 Nov 25. PMID 33234017
- [Background] Farrell SF, Smith AD, Hancock MJ, Webb AL, Sterling M. Cervical spine findings on MRI in people with neck pain compared with pain-free controls: A systematic review and meta-analysis. J Magn Reson Imaging. 2019 Jun;49(6):1638-1654. doi: 10.1002/jmri.26567. Epub 2019 Jan 5. PMID 30614121
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Background] Verhagen AP. Physiotherapy management of neck pain. J Physiother. 2021 Jan;67(1):5-11. doi: 10.1016/j.jphys.2020.12.005. Epub 2020 Dec 24. No abstract available. PMID 33358545
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Corp N, Mansell G, Stynes S, Wynne-Jones G, Morso L, Hill JC, van der Windt DA. Evidence-based treatment recommendations for neck and low back pain across Europe: A systematic review of guidelines. Eur J Pain. 2021 Feb;25(2):275-295. doi: 10.1002/ejp.1679. Epub 2020 Nov 12. PMID 33064878
- [Background] Parikh P, Santaguida P, Macdermid J, Gross A, Eshtiaghi A. Comparison of CPG's for the diagnosis, prognosis and management of non-specific neck pain: a systematic review. BMC Musculoskelet Disord. 2019 Feb 14;20(1):81. doi: 10.1186/s12891-019-2441-3. PMID 30764789
- [Background] Jull GA, Falla D, Vicenzino B, Hodges PW. The effect of therapeutic exercise on activation of the deep cervical flexor muscles in people with chronic neck pain. Man Ther. 2009 Dec;14(6):696-701. doi: 10.1016/j.math.2009.05.004. Epub 2009 Jul 25. PMID 19632880
- [Background] Falla D, Jull G, Hodges P. Training the cervical muscles with prescribed motor tasks does not change muscle activation during a functional activity. Man Ther. 2008 Dec;13(6):507-12. doi: 10.1016/j.math.2007.07.001. Epub 2007 Aug 27. PMID 17720609
- [Background] Villanueva-Ruiz I, Falla D, Lascurain-Aguirrebena I. Effectiveness of Specific Neck Exercise for Nonspecific Neck Pain; Usefulness of Strategies for Patient Selection and Tailored Exercise-A Systematic Review With Meta-Analysis. Phys Ther. 2022 Feb 1;102(2):pzab259. doi: 10.1093/ptj/pzab259. PMID 34935963
- [Background] Fidalgo-Martin I, Ramos-Alvarez JJ, Murias-Lozano R, Rodriguez-Lopez ES. Effects of percutaneous neuromodulation in neuromusculoskeletal pathologies: A systematic review. Medicine (Baltimore). 2022 Oct 14;101(41):e31016. doi: 10.1097/MD.0000000000031016. PMID 36254060
- [Background] Romero-Morales C, Bravo-Aguilar M, Abuin-Porras V, Almazan-Polo J, Calvo-Lobo C, Martinez-Jimenez EM, Lopez-Lopez D, Navarro-Flores E. Current advances and novel research on minimal invasive techniques for musculoskeletal disorders. Dis Mon. 2021 Oct;67(10):101210. doi: 10.1016/j.disamonth.2021.101210. Epub 2021 Jun 4. PMID 34099238
- [Background] Rossi M, DeCarolis G, Liberatoscioli G, Iemma D, Nosella P, Nardi LF. A Novel Mini-invasive Approach to the Treatment of Neuropathic Pain: The PENS Study. Pain Physician. 2016 Jan;19(1):E121-8. PMID 26752480
- [Background] Chakravarthy K, Nava A, Christo PJ, Williams K. Review of Recent Advances in Peripheral Nerve Stimulation (PNS). Curr Pain Headache Rep. 2016 Nov;20(11):60. doi: 10.1007/s11916-016-0590-8. PMID 27671799
- [Derived] Lara-Palomo IC, Romero-Del Rey R, Saavedra-Hernandez M, Garcia-Lopez H, Fernandez-Sanchez M, Cohen SP, Castro-Sanchez AM. Comparison of percutaneous neuromodulation and therapeutic exercise in patients with chronic non-specific neck pain: a study protocol for a randomised controlled trial. BMJ Open. 2025 Jun 12;15(6):e097193. doi: 10.1136/bmjopen-2024-097193. PMID 40506078